CLINICAL TRIAL: NCT05798676
Title: Maternal Characteristics Associated With Child Growth and Adiposity. Search for Nutrigenomic Biomarkers in Peripheral Blood
Brief Title: Maternal Characteristics Associated With Child Growth and Adiposity
Status: Recruiting | Type: Observational
Sponsor: Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri (Other)
Responsible Party: Sponsor
Other Study IDs: L2022
Record Dates: First submitted 2023-02-23; First posted 2023-04-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Obesity, Infant
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Adiposity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and milk
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mothers with pre-pregnancy normal weight and their infants: mothers with pre-pregnancy normal weight according to World Health Organization will provide blood and milk samples
- mothers with pre-pregnancy overweight or obesity and their infants: mothers with pre-pregnancy overweight or obesity according to World Health Organization will provide blood and milk samples
  Interventions: Other: overweight/obesity

INTERVENTIONS:
Other: overweight/obesity — the consequences of maternal pregestational overweight/obesity on infant´s growth and adiposity will be studied
  Groups: mothers with pre-pregnancy overweight or obesity and their infants

SUMMARY:
The goal of this observational study is to investigate the concentrations of leptin, insulin, liver expressed antimicrobial peptide 2 (LEAP2), and cortisol in plasma and breast milk and their relationship with eating behavior, growth, adiposity and with the levels of these hormones in infants, comparing mothers with normal weight and with pre-pregnancy overweight/obesity. The main question[s] it aims to answer are:

* Are maternal hormones associated with child growth and adiposity
* Are maternal hormone receptors associated with child growth and adiposity
* Are infant hormones and their receptors associated with child growth and adiposity
* Are maternal and infant hormones and their receptors associated with child eating behavior Participants will provide milk and blood samples. Researchers will compare mothers with normal weight and with pre-pregnancy overweight/obesity to see if there are differences in child growth and adiposity .

ELIGIBILITY:
Inclusion Criteria:

* Lactating women with pre-pregnancy normal weight and overweight or obesity as described by the World Health Organization.

Exclusion Criteria:

* Diabetes (Type I or II or gestational)
* Multiple pregnancy
* Hypertensive disorders during pregnancy
* Delivery of pre-term infant (<37 weeks).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lactating women with pre-pregnancy normal weight and overweight or obesity recruited at the Mother and Healthy Children Outpatient Service, Instituto de Desarrollo e Investigaciones Pediátricas (IDIP), HIAEP "Sor María Ludovica", La Plata, Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
infant weight | from birth to 2 years old
  weight in kilograms
infant height | from birth to 2 years old
  height in centimeters
infant body mass index (BMI) | from birth to 2 years old
  weight and height will be combined to report BMI in kg/m^2
infant upper arm circumference | from birth to 2 years old
  upper arm circumference in centimeters
infant skinfold thickness | from birth to 2 years old
  skinfold thickness in centimeters
infant blood leptin concentration | six months old
  blood leptin concentration (ng/ml)
infant blood cortisol concentration | six months old
  blood cortisol concentration (ug%)
infant saliva cortisol concentration | six months old
  saliva cortisol (ug%)
infant blood insulin concentration | six months old
  blood insulin concentration (uU/ml)
infant insulin receptor gene expression in peripheral blood mononuclear cells | six months old
  insulin receptor gene expression in peripheral blood mononuclear cells (relative expression)
infant leptin receptor gene expression in peripheral blood mononuclear cells | six months old
  leptin receptor gene expression in peripheral blood mononuclear cells (relative expression)
infant glucocorticoid receptor gene expression in peripheral blood mononuclear cells | six months old
  glucocorticoid receptor gene expression in peripheral blood mononuclear cells (relative expression)
infant blood LEAP2 concentration | six months old
  blood LEAP2 concentration (pg/ml)
infant eating behavior assessed in a Taste acceptance test | at 18 month od
  Outcome Measures Infant taste acceptance was assessed using two complementary measures: an Ingestion Ratio (IR) and a Liking Ratio (LR). Sweet and fat taste acceptance were evaluated using a lactose solution (0.2 M) and a fat emulsion (3.5% w/v), respectively, with water used as a reference. During each test, infants were sequentially offered bottles containing water and the tastant. Intake volume was determined by weighing bottles before and after ingestion.
  The IR was calculated as the volume of tastant consumed divided by the total volume of tastant plus water consumed, allowing comparison across infants by accounting for individual differences in sucking behavior.
  The LR was based on a blinded experimenter's assessment of the infant's overall behavioral response using a standardized 5-point scale ranging from strong rejection to strong acceptance. Both ratios ranged from 0 to 1, with 0.5 indicating indifference relative to water.

SECONDARY OUTCOMES:
maternal blood leptin concentration | 15 days, three and six months postpartum
  blood leptin concentration (ng/ml)
maternal milk leptin concentration | 15 days, three and six months postpartum
  milk leptin concentration (ng/ml)
maternal blood insulin concentration | 15 days, three and six months postpartum
  blood insulin concentration (uU/ml)
maternal milk insulin concentration | 15 days, three and six months postpartum
  milk insulin concentration (uU/ml)
maternal blood cortisol concentration | 15 days, three and six months postpartum
  blood cortisol concentration (ug%)
maternal milk cortisol concentration | 15 days, three and six months postpartum
  milk cortisol concentration (ug%)
maternal insulin receptor gene expression in peripheral blood mononuclear cells | 15 days, three and six months postpartum
  insulin receptor gene expression in peripheral blood mononuclear cells (relative expression)
maternal leptin receptor gene expression in peripheral blood mononuclear cells | 15 days, three and six months postpartum
  leptin receptor gene expression in peripheral blood mononuclear cells (relative expression)
maternal glucocorticoid receptor gene expression in peripheral blood mononuclear cells | 15 days, three and six months postpartum
  glucocorticoid receptor gene expression in peripheral blood mononuclear cells (relative expression)
maternal blood LEAP2 concentration | 15 days, three and six months postpartum
  blood LEAP2 concentration (pg/ml)
maternal milk LEAP2 concentration | 15 days, three and six months postpartum
  milk LEAP2 concentration (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Andreoli, BsC, Principal Investigator — Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri
Locations (1):
- Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri, La Plata, Buenos Aires, Argentina

REFERENCES:
- [Derived] Kruger AL, Malpeli A, Sala M, Casado C, Mendez I, Fotia L, Tournier A, Fasano MV, Andreoli MF. Human milk cortisol is inversely associated with infant BMI and mediates the association between maternal plasma and infant salivary cortisol concentrations. Int J Obes (Lond). 2025 Aug;49(8):1632-1641. doi: 10.1038/s41366-025-01815-4. Epub 2025 May 31. PMID 40450153
- [Derived] Kruger AL, Malpeli A, Sala M, Casado C, Mendez I, Fotia L, Lopez M, Tournier A, Castrogiovanni D, Heredia F, Llovera R, Schioth HB, Perello M, Andreoli MF. The Concentration of Liver-Expressed Antimicrobial Peptide 2 in Human Milk and Infant Plasma Is Positively Associated with Adiposity and Body Weight in the First Year of Life. J Nutr. 2024 Nov;154(11):3388-3399. doi: 10.1016/j.tjnut.2024.09.008. Epub 2024 Sep 12. PMID 39277116